CLINICAL TRIAL: NCT00379288
Title: A 1-Year Safety Study of Medium and High Doses of Mometasone Furoate/Formoterol Combination Formulation and Medium and High Doses of Fluticasone/Salmeterol in Persistent Asthmatics Previously Treated With Medium to High Doses of Inhaled Glucocorticosteroids
Brief Title: Study of Mometasone Furoate/Formoterol Combination and Fluticasone/Salmeterol in Persistent Asthmatics Previously Treated With Inhaled Glucocorticosteroids (P04139)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04139
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Results first posted 2010-08-12 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — BID protein, human; Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MF/F 200/10 mcg BID (Experimental)
  Interventions: Drug: mometasone furoate combination MDI 200/10 mcg BID
- MF/F 400/10 mcg BID (Experimental)
  Interventions: Drug: mometasone furoate combination MDI 400/10 mcg BID
- F/SC 250/50 mcg BID (Active Comparator)
  Interventions: Drug: Fluticasone/Salmeterol 250/50 mcg BID
- F/SC 500/50 mcg BID (Active Comparator)
  Interventions: Drug: Fluticasone/Salmeterol 500/50 mcg BID

INTERVENTIONS:
Drug: mometasone furoate combination MDI 200/10 mcg BID — MF/F 200/10 mcg via a metered dose inhaler (MDI) twice daily for 1 year
  Other Names: SCH 418131
  Arms: MF/F 200/10 mcg BID
Drug: mometasone furoate combination MDI 400/10 mcg BID — MF/F 400/10 mcg via a metered dose inhaler (MDI) twice daily for 1 year
  Other Names: SCH 418131
  Arms: MF/F 400/10 mcg BID
Drug: Fluticasone/Salmeterol 250/50 mcg BID — F/SC 250/50 twice daily for 1 year
  Other Names: Seretide
  Arms: F/SC 250/50 mcg BID
Drug: Fluticasone/Salmeterol 500/50 mcg BID — F/SC 500/50 twice daily for 1 year
  Other Names: Seretide
  Arms: F/SC 500/50 mcg BID

SUMMARY:
The purpose of this study is to evaluate the long-term safety of mometasone furoate/formoterol (MF/F) metered dose inhaler (MDI) 200/10 mcg twice-a-day (BID) and MF/F MDI 400/10 mcg BID and two doses of fluticasone/salmeterol combination (F/SC) (250/50 mcg BID and 500/50 mcg BID) in subjects with persistent asthma who require maintenance treatment on inhaled glucocorticosteroids (ICS); evaluator-blind.

In addition, the extrapulmonary effects on 24-hour plasma cortisol area under curve (AUC), of MF/F MDI 200/10 mcg BID, MF/F MDI 400/10 mcg BID, F/SC MDI 250/50 mcg BID, and F/SC MDI 500/50 mcg BID will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either sex and any race, at least 12 years of age, with a diagnosis of asthma of at least 12 months.
* Use of medium or high daily dose of ICS (alone or in combination with long-acting beta-agonist [LABA]) for at least 12 weeks prior to Screening and have been on a stable regimen for at least 2 weeks prior to Screening.

  * Medium daily doses of ICS:

    * > 500 to 1000 mcg beclomethasone chlorofluorocarbon (CFC)
    * > 250 to 500 mcg beclomethasone hydrofluoroalkane (HFA)
    * > 600 to 1000 mcg budesonide dry powder inhaler (DPI)
    * > 1000 to 2000 mcg flunisolide
    * > 250 to 500 mcg fluticasone
    * 400 mcg MF
    * > 1000 to 2000 mcg triamcinolone acetonide
  * High daily doses of ICS:

    * > 1000 mcg beclomethasone CFC
    * > 500 mcg beclomethasone HFA
    * > 1000 mcg budesonide DPI
    * > 2000 mcg flunisolide
    * > 500 mcg fluticasone
    * > 400 mcg MF
    * > 2000 mcg triamcinolone acetonide
* If there is no inherent harm in changing the subject's current asthma therapy, the subject must discontinue prescribed ICS or ICS/LABA combination at Baseline.
* Must show evidence of reversibility within the last 12 months or during the Screening Period. Historical reversibility defined as an increase in absolute forced expiratory volume in 1 second (FEV1) of >= 12% and >= 200 mL will qualify if performed within 12 months of Screening. If no historical reversibility, subject must demonstrate an absolute FEV1 of >= 12% and >= 200 mL within 10 to 15 minutes after four puffs of salbutamol at Visit 1 or anytime prior to Baseline.
* At Screening and Baseline, FEV1 must be >= 50% predicted, when restricted medications are withheld for the appropriate intervals.
* Complete blood count, blood chemistries, urinalysis, and electrocardiogram (ECG) conducted at Screening must be within normal limits or clinically acceptable to the investigator/sponsor. A chest x-ray performed at Screening or within 12 months prior must be clinically acceptable.
* A female of childbearing potential must be using a medically acceptable, adequate form of birth control:

  * prescribed hormonal contraceptives;
  * medically prescribed intrauterine device (IUD);
  * medically prescribed transdermal contraceptive;
  * condom in combination with spermicide;
  * monogamous relationship with a male partner who has had a vasectomy.

Birth control must have started at least 3 months prior to Screening. Subject must agree to continue its use for the duration of the study. A subject of childbearing potential who is not currently sexually active must agree to use a medically acceptable method should she become sexually active during the study. Women who have been surgically sterilized or are at least 1 year postmenopausal are not considered to be of childbearing potential. A subject of childbearing potential must have a negative serum pregnancy test at Screening.

Key Exclusion Criteria:

* A change (increase or decrease) in absolute FEV1 of > 20% at any time from the Screening Visit up to, and including, the Baseline Visit.
* A subject who requires the use of > 12 inhalations per day of short-acting beta-agonist (SABA) MDI or > 2 nebulized treatments per day of 2.5 mg salbutamol, on any 2 consecutive days from the Screening Visit up to, and including, the Baseline Visit.
* A subject who experiences a clinical asthma exacerbation (defined as a deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication [other than SABA]) at any time from the Screening Visit up to, and including, the Baseline Visit.
* A subject who has ever required ventilator support for respiratory failure secondary to asthma.
* A subject who is a smoker or ex-smoker and has smoked within the previous year or has had a cumulative smoking history > 10 pack-years.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maspero JF, Nolte H, Cherrez-Ojeda I; P04139 Study Group. Long-term safety of mometasone furoate/formoterol combination for treatment of patients with persistent asthma. J Asthma. 2010 Dec;47(10):1106-15. doi: 10.3109/02770903.2010.514634. Epub 2010 Nov 1. PMID 20874458
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Maspero J, Cherrez I, Doherty DE, Tashkin DP, Kuna P, Kuo WL, Gates D, Nolte H, Chylack LT Jr. Appraisal of lens opacity with mometasone furoate/formoterol fumarate combination in patients with COPD or asthma. Respir Med. 2014 Sep;108(9):1355-62. doi: 10.1016/j.rmed.2014.04.015. Epub 2014 May 2. PMID 25044280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects starting study are those subjects who completed screening procedures and randomized.
Groups:
- MF/F 200/10 mcg BID: mometasone furoate/formoterol (MF/F) 200/10 mcg via a metered dose inhaler (MDI) twice daily for 1 year
- MF/F 400/10 mcg BID: MF/F 400/10 mcg via a metered dose inhaler (MDI) twice daily for 1 year
- F/SC 250/50 mcg BID: fluticasone/salmeterol combination (F/SC) 250/50 twice daily for 1 year
- F/SC 500/50 mcg BID: F/SC 500/50 twice daily for 1 year
Period: Overall Study
Arm/Group | MF/F 200/10 mcg BID | MF/F 400/10 mcg BID | F/SC 250/50 mcg BID | F/SC 500/50 mcg BID
Started | 141 | 130 | 68 | 65
Completed | 122 | 108 | 58 | 57
Not Completed | 19 | 22 | 10 | 8
Not completed — Adverse Event | 5 | 6 | 2 | 0
Not completed — Treatment Failure | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 3 | 3 | 2 | 0
Not completed — Subject withdrew-unrelated to study drug | 0 | 3 | 4 | 2
Not completed — Subject withdrew-related to study drug | 1 | 0 | 0 | 1
Not completed — Noncompliance with protocol | 8 | 6 | 2 | 1
Not completed — Did not meet protocol eligibility | 0 | 1 | 0 | 2
Not completed — Administrative | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MF/F 200/10 mcg BID: MF/F 200/10 mcg via a metered dose inhaler (MDI) twice daily for 1 year
- F/SC 250/50 mcg BID: F/SC 250/50 twice daily for 1 year
- Total: Total of all reporting groups
Arm/Group | MF/F 200/10 mcg BID | MF/F 400/10 mcg BID | F/SC 250/50 mcg BID | F/SC 500/50 mcg BID | Total
Number analyzed (Participants) | 141 | 130 | 68 | 65 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (15.2) | 39.3 (14.5) | 32.4 (14.9) | 37.1 (15.0) | 35.5 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 86 | 38 | 40 | 256
  Male | 49 | 44 | 30 | 25 | 148

OUTCOME MEASURES:

1. Primary Outcome: The Number of All Randomized Subjects Reporting Adverse Events (AEs).
Description: AEs that are considered Related, Severe, and Serious, as determined by the investigator and using specific criteria defined in the protocol, are included in the primary results.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | MF/F 200/10 mcg BID | MF/F 400/10 mcg BID | F/SC 250/50 mcg BID | F/SC 500/50 mcg BID
Number analyzed (Participants) | 141 | 130 | 68 | 65
participants
  Treatment-Emergent Adverse Events (TEAE) | 109 | 103 | 56 | 50
  Related Adverse Events | 40 | 30 | 16 | 13
  Severe Adverse Events | 8 | 5 | 4 | 4
  Serious Adverse Events | 7 | 8 | 4 | 2
Statistical Analysis 1: Comparison: MF/F 200/10 mcg BID; Test type: Superiority or Other; percentage of subjects with TEAEs = 77.4
Statistical Analysis 2: Comparison: MF/F 200/10 mcg BID; Test type: Superiority or Other; percentage of subjects with related AEs = 28.4
Statistical Analysis 3: Comparison: MF/F 200/10 mcg BID; Test type: Superiority or Other; percentage of subjects with severe AEs = 5.7
Statistical Analysis 4: Comparison: MF/F 200/10 mcg BID; Test type: Superiority or Other; percentage of subjects with serious AEs = 4.9
Statistical Analysis 5: Comparison: MF/F 400/10 mcg BID; Test type: Superiority or Other; percentage of subjects with TEAEs = 79.2
Statistical Analysis 6: Comparison: MF/F 400/10 mcg BID; Test type: Superiority or Other; percentage of subjects with related AEs = 23.1
Statistical Analysis 7: Comparison: MF/F 400/10 mcg BID; Test type: Superiority or Other; percentage of subjects with severe AEs = 3.8
Statistical Analysis 8: Comparison: MF/F 400/10 mcg BID; Test type: Superiority or Other; percentage of subjects with serious AEs = 6.1
Statistical Analysis 9: Comparison: F/SC 250/50 mcg BID; Test type: Superiority or Other; percentage of subjects with TEAEs = 82.4
Statistical Analysis 10: Comparison: F/SC 250/50 mcg BID; Test type: Superiority or Other; percentage of subjects with related AEs = 23.5
Statistical Analysis 11: Comparison: F/SC 250/50 mcg BID; Test type: Superiority or Other; percentage of subjects with severe AEs = 5.9
Statistical Analysis 12: Comparison: F/SC 250/50 mcg BID; Test type: Superiority or Other; percentage of subjects with serious AEs = 5.8
Statistical Analysis 13: Comparison: F/SC 500/50 mcg BID; Test type: Superiority or Other; percentage of subjects with TEAEs = 76.9
Statistical Analysis 14: Comparison: F/SC 500/50 mcg BID; Test type: Superiority or Other; percentage of subjects with related AEs = 20
Statistical Analysis 15: Comparison: F/SC 500/50 mcg BID; Test type: Superiority or Other; percentage of subjects with severe AEs = 6.2
Statistical Analysis 16: Comparison: F/SC 500/50 mcg BID; Test type: Superiority or Other; percentage of subjects with serious AEs = 3.1

ADVERSE EVENTS:
Groups:
- MF/F MDI 200/10 mcg BID: MF/F 200/10 mcg via a metered dose inhaler (MDI) twice daily for 1 year
- MF/F MDI 400/10 mcg BID: MF/F 400/10 mcg via a metered dose inhaler (MDI) twice daily for 1 year
- F/SC MDI 250/50 mcg BID: F/SC 250/50 twice daily for 1 year
- F/SC MDI 500/50 mcg BID: F/SC 500/50 twice daily for 1 year
Arm/Group | MF/F MDI 200/10 mcg BID | MF/F MDI 400/10 mcg BID | F/SC MDI 250/50 mcg BID | F/SC MDI 500/50 mcg BID
Serious Adverse Events (participants affected / at risk) | 7/141 | 8/130 | 4/68 | 2/65
Other Adverse Events (participants affected / at risk) | 93/141 | 82/130 | 51/68 | 41/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 200/10 mcg BID (N=141) | MF/F MDI 400/10 mcg BID (N=130) | F/SC MDI 250/50 mcg BID (N=68) | F/SC MDI 500/50 mcg BID (N=65)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LENS DISORDER (Eye disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
OCULAR HYPERTENSION (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELECTROCUTION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTEBRAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 200/10 mcg BID (N=141) | MF/F MDI 400/10 mcg BID (N=130) | F/SC MDI 250/50 mcg BID (N=68) | F/SC MDI 500/50 mcg BID (N=65)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 6 (9) | 3 (4) | 5 (6)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (7) | 7 (10) | 3 (8) | 3 (3)
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 3 (5) | 3 (4) | 4 (4) | 0 (0)
PYREXIA (General disorders) | 8 (11) | 6 (6) | 4 (5) | 1 (2)
BRONCHITIS (Infections and infestations) | 17 (23) | 20 (29) | 14 (17) | 7 (7)
INFLUENZA (Infections and infestations) | 14 (23) | 13 (16) | 9 (13) | 11 (13)
NASOPHARYNGITIS (Infections and infestations) | 29 (39) | 21 (34) | 13 (19) | 8 (9)
PHARYNGITIS (Infections and infestations) | 15 (24) | 11 (11) | 9 (12) | 9 (9)
RHINITIS (Infections and infestations) | 7 (10) | 7 (7) | 8 (9) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (6) | 5 (9) | 5 (5) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (13) | 6 (8) | 7 (11) | 3 (3)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (8) | 2 (6) | 4 (7)
HEADACHE (Nervous system disorders) | 33 (77) | 31 (85) | 17 (47) | 13 (31)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 2 (5) | 4 (4) | 2 (2)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 7 (25) | 5 (9) | 5 (5) | 2 (2)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 11 (20) | 7 (10) | 2 (3) | 1 (1)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 11 (24) | 9 (18) | 6 (11) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish/present any interim results without prior sponsor written consent. The investigator agrees to provide to the sponsor, 45 days prior to submission, review copies for publication that report any study results. The sponsor has the right to review and comment. If the parties disagree, investigator agrees to meet with the sponsor, prior to submission for publication, to discuss and resolve any such issues/disagreement.